CLINICAL TRIAL: NCT00455728
Title: International Cooperative Growth Study (iNCGS) Post Marketing Surveillance Program for NutropinAq® [Somatropin (rDNA Origin) Injection]
Brief Title: A Post Marketing Surveillance Program for NutropinAq® in Paediatric Growth Disorders
Acronym: iNCGS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 2-79-58035-005; EUPAS7948 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Growth Hormone Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a multicenter, open label, observational, post marketing surveillance study of NutropinAq® in Austria, France, Germany, Italy, Spain, Romania and United Kingdom to collect long-term safety and effectiveness information on NutropinAq® during treatment of paediatric growth disorders.

DETAILED DESCRIPTION:
The objective of this study is to collect long term safety and effectiveness information on Ipsen's growth hormone (GH) NutropinAq® regarding treatment of paediatric growth disorders for which GH is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex who are treated with NutropinAq® for the treatment of growth failure
* Patients who are willing to comply with follow-up appointments throughout study participation
* Written informed consent signed by both parents or by the liable parent or by the legal guardian when applicable, and by the child when applicable

Exclusion Criteria:

* Patients not treated with NutropinAq®
* Patients with closed epiphyses
* Patients with active neoplasia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children treated with NutropinAq in the specialised paediatric endocrinology centres
Sampling Method: Non-Probability Sample
Enrollment: 3690 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Every 3 months until study completion
  Description and incidence of any Serious Adverse Event (SAE) and all related (serious and non-serious) Adverse Events (AEs).

SECONDARY OUTCOMES:
Treatment height measurements until epiphyseal closure is achieved. | Every 3 months until study completion

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Slough, Berkshire, United Kingdom

REFERENCES:
- [Derived] Coutant R, Bosch Munoz J, Dumitrescu CP, Schnabel D, Sert C, Perrot V, Dattani M. Effectiveness and Overall Safety of NutropinAq(R) for Growth Hormone Deficiency and Other Paediatric Growth Hormone Disorders: Completion of the International Cooperative Growth Study, NutropinAq(R) European Registry (iNCGS). Front Endocrinol (Lausanne). 2021 May 25;12:676083. doi: 10.3389/fendo.2021.676083. eCollection 2021. PMID 34113318